CLINICAL TRIAL: NCT05888038
Title: Virtual Reality's Effect on Decreasing Pain and Subsequent Opioid Use in Pediatric Patients in the Post-Operative Period Following Scoliosis Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-0286
Record Dates: First submitted 2022-09-03; First posted 2023-06-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Scoliosis; Juvenile; Scoliosis; Adolescence; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention - use of VR (Experimental)
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — virtual reality

SUMMARY:
The goal of this study is to determine whether introducing VR in the immediate post-operative period following scoliosis repair can reduce perceived pain and stress in pediatric patients and in turn ultimately decrease opioid use. Based on previous studies that have been performed in other fields of pediatrics showing a decrease in pain and stress with VR use, the investigators hypothesize that VR will significantly decrease patient's reported level of pain and stress immediately following the VR session, and that patients will require less opioids during their inpatient stay as a result.

DETAILED DESCRIPTION:
This project evaluates whether providing pediatric post-operative scoliosis repair patients with a virtual reality (VR) session at specific time point following surgery can decrease pain and stress experienced and if this leads to a decrease in the use of pain medications required during the immediate recovery period. Virtual reality technology was ordered to use as a distraction tool as part of routine pediatric care for hospitalized patients. The study involves measuring pain and stress using validated scales as well as calculating opioid use in this specific pediatric post-operative scoliosis repair population. All post-operative scoliosis repair patients admitted to the inpatient pediatric floor above 7 years of age will be eligible for participation in this study. The goal is to collect data on at least 50 patients over the course of 12-18 months. Parental consent and child assent will be obtained on day 2 post-op surgery using a standardized consent and assent form, respectively. Data will be collected from the Numerical Pain Rating Scale and the State Trait Anxiety Inventory, which will be administered pre- and post-VR sessions, with the goal of comparing scores to evaluate for any decrease in pain and stress levels. Data on inpatient opioid use post-operatively will be used to compare with previous post-operative scoliosis patients to determine whether there a significant decrease in opioid use in the subjects exposed to VR. During the data collection process, results will be documented in an organized but deidentified manner.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients post scoliosis repair
* age 7-21

Exclusion Criteria:

* age less than 7 years;
* history of seizures, epilepsy,
* history of motion sickness/balance problems,
* susceptibility to migraines
* currently pregnant

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | 2 years
  Use of virtual reality device exercise to reduce perception of pain. Participant will complete Numerical Pain Rating Scale.
Stress Assessment | 2 years
  Participant will complete and the State Trait Anxiety Inventory to assess stress

CONTACTS AND LOCATIONS:
Locations (1):
- SIUH Northwell Health, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No